CLINICAL TRIAL: NCT00174577
Title: Risperidone Augmentation Therapy in Patients Who Have Failed or Only Partially Responded to an Adequate Trial of Antidepressant
Brief Title: Risperidone Augmentation Therapy in Patients Who Have Failed or Only Partially Responded to a Trial of Antidepressant
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rhode Island Hospital (Other)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry); Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIS-Dep-402
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
The purpose of this study is to assess the safety and efficacy of risperidone augmentation in patients who have failed to respond or only partially responded to an adequate trial of an antidepressant.

DETAILED DESCRIPTION:
Specific Aims: The goal of this study was to assess the safety and efficacy of risperidone augmentation in patients with major depression who failed to respond, or only partially responded, to an adequate trial of an antidepressant medication. Patients who met this criteria received adjunctive risperidone (1- 3 mg.) for an additional four-week treatment trial.

Subject Population: A total sample of 84 patients completed the study at two sites (Rhode Island Hospital/Brown University, n=42, Emory University, n=42).

Methods/Design: Patients who met criteria for unipolar depression and failed to respond, or partially responded, to an adequate trial of antidepressant medication were randomized to risperidone or a placebo for an additional 4 week treatment trial while continuing on the same dose of their antidepressant medication. Randomization was at a 2:1 ratio of risperidone to placebo.

Data Analysis: Patient outcome (recovery status) of the two treatment conditions were compared using a MADRS rating < 10 to denote remission while improvement was defined as a 50% decrease from baseline to end of study. Odds ratio were examined to see if risperidone augmentation significantly affected the chance of recovery from depression at the end of 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with major depression or partially remitted depression
* currently receiving an adequate trial of an antidepressant

Exclusion Criteria:

* diagnosis of bipolar I or bipolar II disorder
* psychotic features
* substance dependence or abuse in the past three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84
Dates: Start 2003-02; Study Completion 2005-02

PRIMARY OUTCOMES:
Depression symptoms,change score on MADRS scale at 4 weeks
Group differences on HRS-D scores
Group differences on remission and improvement

SECONDARY OUTCOMES:
Between group differences on quality-of-life measures
Group differences of anxiety and psychosocial factors

CONTACTS AND LOCATIONS:
Overall Officials: Gabor I Keitner, M.D., Principal Investigator — Rhode Island Hospital/Brown University
Locations (2):
- United States (2):
  - Emory University School of Medicine, Atlanta, Georgia
  - Mood Disorders Program - Rhode Island Hospital, Providence, Rhode Island